CLINICAL TRIAL: NCT01137955
Title: Double-blind Randomized Controlled Trial of Rifaximin for Persistent Symptoms in Patients With Celiac Disease
Brief Title: Rifaximin for the Treatment of Persistent Symptoms in Patients With Celiac Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAB6531; IRB-AAAB6531(Y3M00) (Other: Columbia University Medical Center IRB)
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Celiac Disease
Keywords: Gastrointestinal Symptom Rating Scale (GSRS); Poorly responsive; Refractory; Small intestine bacterial overgrowth; Breath test
MeSH Terms: conditions — Celiac Disease | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rifaximin 400mg (Experimental): Antibiotic ,Rifaximin 400mg, given 3 times a day for 10 days.
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator): Placebo pills given 3 times a day for 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — Rifaximin 400mg orally three times a day for 10 days total
  Other Names: Placebo orally three times a day for 10 days total
  Arms: Rifaximin 400mg
Drug: Placebo — Placebo orally three times a day for 10 days total
  Other Names: Rifaximin 400 mg orally three times a day for 10 days total
  Arms: Placebo

SUMMARY:
Celiac disease is a condition in which the small intestine is damaged by gluten, the storage protein of wheat and similar proteins in barley and rye. The disease can cause different symptoms such as diarrhea, bloating, abdominal pain and weight loss. The majority of patients respond to a gluten-free diet. However some patients (5-30%) have persistent symptoms and are considered to be poor responders to the diet. Bacterial overgrowth in the small intestine accounts for some of the refractory patients.

This study seeks to determine if antibiotic therapy with rifaximin relieves the symptoms of patients who are poorly responsive to a gluten-free diet and whether this impacts their breath test results.

DETAILED DESCRIPTION:
A symptom questionnaire will be administered at study initiation, 2 weeks and 12 weeks. Patients will undergo a breath test which involves drinking a sugar (lactulose) solution and breathing into a machine. This technique will identify the presence of bacteria in the small intestine. They will be randomly selected to receive either an antibiotic (rifaximin) or placebo three times a day for 10 days to treat their bacterial overgrowth.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age 18 or older
* Biopsy proven celiac disease
* Persistent symptoms of diarrhea, gas, bloating and/or cramping despite a gluten free diet for at least 1 month
* Women that are not pregnant or lactating can be included. All women must have a documented negative pregnancy test at the initiation of the study. Women who become pregnant during the study will be asked to discontinue the study drug and will be followed up until the outcome of pregnancy is known. Women of child bearing potential must be practicing an effective method of birth control (eg: prescription oral contraceptive, contraceptive injections, intra-uterine device (IUD), double barrier method, contraceptive patch, male sterilization) before entry and throughout the treatment period.

Exclusion Criteria:

1. antibiotic use for any indication within preceding one month
2. use of bismuth compounds within preceding month
3. concomitant use of pancreatic supplements
4. concomitant use of antispasmodics
5. concomitant use of immunomodulators such as corticosteroids, budesonide, alkylating agents and antimetabolites.
6. concomitant use of probiotics
7. concomitant use of prokinetic agents
8. concomitant use of 5-hydroxytryptamine receptor (5HT3) antagonists,5-hydroxytryptamine receptor (5HT4) antagonists.
9. concomitant use of antimotility agents (e.g loperamide)
10. concomitant use of antidiarrheal agents
11. diagnosed microscopic colitis or inflammatory bowel disease
12. other causes of malabsorption: pancreatic insufficiency, giardiasis and enteropathy associated with T cell lymphoma.
13. other diseases: renal or hepatic insufficiency.
14. pregnant patients and lactating females. In addition women of child bearing age will be excluded if they are not using one of the methods of contraception like oral contraceptives,intrauterine device.

    and double barrier methods.
15. patients with tuberculosis or a positive purified protein derivative (PPD) test and infection with other mycobacterial diseases.
16. allergy and/or potential emergence of drug resistance to rifampicin and rifamycin compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter HR Green, MD, Principal Investigator — Columbia University
Locations (1):
- Celiac Disease Center at Columbia University, New York, New York, United States

REFERENCES:
- [Result] Chang MS, Minaya MT, Cheng J, Connor BA, Lewis SK, Green PH. Double-blind randomized controlled trial of rifaximin for persistent symptoms in patients with celiac disease. Dig Dis Sci. 2011 Oct;56(10):2939-46. doi: 10.1007/s10620-011-1719-6. Epub 2011 Jun 7. PMID 21647654

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from Celiac Disease Center.
Pre-assignment Details: Fifty participants were enrolled and 41 participants completed the trial.
Groups:
- Rifaximin: Antibiotic ( 25 subjects)
  400 mg capsules of Rifaximin 3 times a day for 10 days.
- Placebo: Inert capsules ( 25 Subjects)
  Placebo capsules 3 times a day for 10 days.
Period: Overall Study
Arm/Group | Rifaximin | Placebo
Started | 25 | 25
Completed | 20 | 21
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifaximin | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (14.6) | 43.4 (14.0) | 42.7 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Baseline Gastrointestinal Symptom Rating Scale (GSRS) Score
Description: Validated seven point questionnaire that assesses gastrointestinal symptoms for five symptom areas, including abdominal pain, reflux, indigestion, diarrhea, and constipation. Individual scores are calculated for each symptom area and the mean of the scores is used to derive an overall GSRS score. Scores range from 0-7, with higher scores indicating gastrointestinal discomfort.
Time Frame: Baseline (week 0)
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Rifaximin: 400 mg capsules of Rifaximin 3 times a day for 10 days.
- Placebo: Placebo capsules 3 times a day for 10 days.
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 20 | 21
Score on a scale | 2.7 (1.1) | 2.8 (0.9)

2. Primary Outcome: Week 2 Gastrointestinal Symptom Rating Scale (GSRS) Score
Description: as for outcome 1
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Rifaximin 400mg: 400 mg capsules of Rifaximin 3 times a day for 10 days.
Arm/Group | Rifaximin 400mg | Placebo
Number analyzed (Participants) | 20 | 21
score on a scale | 2.3 (0.6) | 2.4 (0.6)

3. Secondary Outcome: Percentage of Participants With Abnormal Breath Test
Description: A breath test measures for small intestine bacterial overgrowth (SIBO). The breath test measures the amount of hydrogen exhaled after drinking a sugar (lactulose) solution. An abnormal breath test is defined as: 1) a rise in hydrogen of ≥20 parts per million (ppm) within 100 minutes, or 2) two peaks ≥20 ppm over baseline.
Time Frame: Up to 12 weeks
Measure: Number; unit: Percent of Participants
Arm/Group | Rifaximin | Placebo
Number analyzed (Participants) | 20 | 21
Percent of Participants | 12 | 20

4. Primary Outcome: Week 12 Gastrointestinal Symptom Rating Scale (GSRS) Score
Description: as for outcome 1
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rifaximin 400mg | Placebo
Number analyzed (Participants) | 20 | 21
score on a scale | 2.5 (0.8) | 2.5 (0.8)

ADVERSE EVENTS:
Groups:
- Rifaximin: Antibiotic: Rifaximin 400mg orally three times a day for 10 days total
- Placebo: Inert capsules: Placebo orally three times a day for 10 days total
Arm/Group | Rifaximin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

LIMITATIONS AND CAVEATS:
Small sample size. Challenges of diagnosing bacterial overgrowth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No